CLINICAL TRIAL: NCT04446767
Title: Photobiomodulation With Polarized Light as Adjunctive Treatment in Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Taha, ASSISTANT PROFESSOR, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T REC/017/00482.
Record Dates: First submitted 2020-05-28; First posted 2020-06-25 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Wound Healing Disorder
Keywords: diabetes; foot ulcer; polarized light; ;wound healing
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer | interventions — Microscopy, Polarization

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioptron light therapy and medical care (Experimental): bioptron light therapy sessions, about 12 minutes on the foot ulcer 3 sessions per week for about 8 weeks plus medical care in the form of Appropriate day-care and principles of local ulcer therapy, washing and bandaging, use of anti exudative, anti-inflammatory and disinfection solutions will be administered to this group, topical antibiotics will be administered based on bio-gram and antibiogram results
  Interventions: Radiation: polarized light
- medical care (Active Comparator): Appropriate day-care and principles of local ulcer therapy, washing and bandaging, use of anti exudative, anti-inflammatory and disinfection solutions will be administered to this group, topical antibiotics will be administered based on bio-gram and antibiogram results
  Interventions: Other: Medical Care

INTERVENTIONS:
Radiation: polarized light — bioptron light therapy sessions, about 12 minutes on the foot ulcer 3 sessions per week for about 8 weeks
  Other Names: bioptron light therapy
  Arms: Bioptron light therapy and medical care
Other: Medical Care — Appropriate day-care and principles of local ulcer therapy, washing and bandaging, use of anti exudative, anti-inflammatory and disinfection solutions will be administered to this group, topical antibiotics will be administered based on bio-gram and antibiogram results
  Arms: medical care

SUMMARY:
Effect of Photobiomodulation With Polarized Light on wound healing and aerobic microflora in Diabetic Foot Ulcer

DETAILED DESCRIPTION:
Effect of Photobiomodulation With Polarized Light on wound healing and aerobic microflora in Diabetic Foot Ulcer both sexes were included and intervention will be given for two months, wound healing will be assessed by measuring the surface area and the Aerobic microflora will be isolated and controlled on the basis of bio-gram and antibiogram at the beginning and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with diagnosed diabetic foot ulcer lasting at least 4 weeks ( sized from 0.5 to 2 cm
2. Cooperative and mentally stable patients .

Exclusion Criteria:

1. Hepatic patients .
2. Uncontrolled hypertension .
3. Uncontrolled diabetic patients with HbA1c>8.5% .
4. Neurological disorders .
5. Musculoskeletal disorders that interfere with program .
6. Previous history or any sign of DVT .

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Histologic evaluation: | two months
  Aerobic microflora will be isolated and controlled on the basis of biogram and antibiogram at the beginning and at the end of treatment
Wound assessment | two months
  The wound surface area (ulcer size), lenghth and width will measured using Ruler technique

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taha MM, El-Nagar MM, Elrefaey BH, Elkholy RM, Ali OI, Alkhamees N, Felaya EEE. Effect of Polarized Light Therapy (Bioptron) on Wound Healing and Microbiota in Diabetic Foot Ulcer: A Randomized Controlled Trial. Photobiomodul Photomed Laser Surg. 2022 Dec;40(12):792-799. doi: 10.1089/photob.2021.0175. Epub 2022 Oct 28. PMID 36315226